CLINICAL TRIAL: NCT03590054
Title: A Phase 1b Dose Escalation/Expansion Study of Abexinostat in Combination With Pembrolizumab in Patients With Advanced Solid Tumor Malignancies
Brief Title: Abexinostat in Combination With Pembrolizumab in Patients With Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rahul Aggarwal (Other)
Collaborators: Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Assistant Professor of Hematology/Oncology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18956; NCI-2018-01395 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Stage III Cutaneous Melanoma; Stage IV Cutaneous Melanoma; Locally Advanced Melanoma; Locally Advanced Solid Neoplasm; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Urothelial Carcinoma; Non-Small Cell Lung Carcinoma; Stage IB Lung Cancer AJCC v7; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Ureteral Neoplasms | interventions — abexinostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation: (abexinostat, pembrolizumab) (Experimental): Participants receive abexinostat PO BID on days -7 to -4 of the lead-in period, and days 1-4, 8-11 of each treatment cycle and pembrolizumab over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abexinostat; Biological: Pembrolizumab
- Cohort A: Dose Expansion (abexinostat, pembrolizumab) (Experimental): Participants with primary resistance to prior anti-PD-1/PD-L1 will receive abexinostat PO BID on days -7 to -4 of the lead-in period, and days 1-4, 8-11 of each treatment cycle and pembrolizumab over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abexinostat; Biological: Pembrolizumab
- Cohort B: Dose Expansion (abexinostat, pembrolizumab) (Experimental): Participants with acquired resistance, defined as treatment duration on prior CPI for greater than 6 months with evidence of clinical benefit (tumor regression or disease stabilization) with subsequent disease progression will receive abexinostat PO BID on days -7 to -4 of the lead-in period, and days 1-4, 8-11 of each treatment cycle and pembrolizumab over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abexinostat; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Abexinostat — Given orally (PO) twice a day (BID) days 1-4, 8-11 of every 21 day cycle
  Other Names: PCI-24781
Biological: Pembrolizumab — Given IV on day 1 of every 21 day cycle
  Other Names: Keytruda

SUMMARY:
This phase I trial studies the best dose and side effects of abexinostat and how well it works with given together with pembrolizumab in treating participants with microsatellite instability (MSI) solid tumors that have spread to other places in the body. Abexinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Giving abexinostat and pembrolizumab may work better in treating participants with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated and recommended phase 2 dose of abexinostat in combination with anti-PD-1/PD-L1 checkpoint inhibitor (CPI). (Dose escalation)

II. To determine the objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in patients treated with abexinostat in combination with CPI in patients with prior primary (cohort A) or acquired (cohort B) resistance to prior CPI treatment. (Dose expansion)

SECONDARY OBJECTIVES:

I. To determine the objective response rate and median duration of response (DoR) by immune modified (i)RECIST criteria.

II. To determine the median progression-free survival (PFS).

III. To further characterize the safety profile of the treatment combination.

OUTLINE: This is a dose-escalation study of abexinostat.

Participants receive abexinostat orally (PO) twice daily (BID) on days 1-21 and pembrolizumab intravenously (IV) on over 30 minutes day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient >= 18 years of age at the time of study enrollment.
* Has histologically confirmed locally advanced or metastatic solid tumor malignancy with one of the following tumor types:

  * Urothelial carcinoma
  * Melanoma
  * Non-small cell lung cancer
  * Small cell lung cancer
  * Non-pulmonary squamous cell carcinoma
  * Head and neck squamous cell carcinoma
  * MSI-high solid tumor, with MSI-high status defined by microsatellite instability testing by Polymerase chain reaction (PCR), loss of mismatch repair proteins by Immunohistochemistry (IHC), or Clinical Laboratory Improvement Amendments (CLIA)-approved next generation sequencing test.
  * Gastric and gastro-esophageal junction adenocarcinoma
  * Merkel cell carcinoma
  * Thymic carcinoma
  * Mesothelioma
* Measurable disease by RECIST 1.1 criteria.
* Dose Expansion only:

  * Disease progression during or within 3 months of last dose of most recent line of prior anti-PD-1/PD-L1-based treatment with a pattern of progression as defined as one of the following:

    * Primary Resistance (Cohort A): Progressive disease as best response to prior treatment with anti-PD-1/PD-L1 treatment
    * Acquired Resistance (Cohort B): Stable disease, partial response or complete response to prior anti-PD-1/PD-L1 treatment with subsequent disease progression during or within 3 months following last dose of anti-PD-1/PD-L1 treatment
  * A tumor biopsy is mandatory unless

    * There is no safely accessible lesion, OR
    * Archival metastatic tumor tissue is available with sufficient quantity that was obtained following the last dose of most recent systemic therapy.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Has adequate baseline organ function, as demonstrated by the following:

  * Serum creatinine =< 1.5 x institutional upper limit of normal (ULN) or calculated creatinine clearance > 50 mL/min
  * Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN (patients with hepatic metastases must have AST/ALT =< 5 x ULN).
  * Absolute neutrophil count (ANC) >= 1.5 x 10^9/L.
  * Hemoglobin >= 8 g/dL.
  * Platelet count >= 75 x 10^9/L.
* Agrees to use acceptable contraceptive methods for the duration of time on the study, and continue to use acceptable contraceptive methods for 6 months (after the last treatment with study treatment.
* Has provided signed informed consent before initiation of any study-specific procedures or treatment.
* Men treated or enrolled on this protocol must agree to use adequate contraception the duration of study participation and 3 months after completion of study drug administration.

Exclusion Criteria:

* Has persistent clinically significant toxicities (grade >= 2; per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5) from previous anticancer therapy (excluding alopecia which is permitted and excluding grades 2 and 3 laboratory abnormalities if they are not associated with symptoms, are not considered clinically significant by the Investigator, and can be managed with available medical therapies).
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/ interstitial lung disease
* Has a diagnosis of clinically significant immunodeficiency.
* Has received external-beam radiation or another systemic anticancer therapy within 14 days or 5 half-lives (whichever is shorter) before start of study treatment.
* Has received treatment with an investigational drug or monoclonal antibody within 28 days prior to study treatment administration. For classes of investigational agents that are not known to have prolonged toxicities, the washout time may be decreased to 14 days at the discretion of the principal investigator.
* Has received previous treatment with a histone deacetylase (HDAC) inhibitor.
* Has an additional active malignancy that may confound the assessment of the study endpoints. Patients with the following concomitant neoplastic diagnoses are eligible: nonmelanoma skin cancer and carcinoma in situ including transitional cell carcinoma, anal carcinoma, and melanoma in situ).
* Has clinically significant cardiovascular disease including, but not limited to:

  * Uncontrolled or any New York Heart Association class 3 or 4 congestive heart failure
  * Uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months before study entry
  * Clinically significant arrhythmias not controlled by medication.
* Has a history of untreated brain, or leptomeningeal, metastases (central nervous system (CNS) imaging is not required before study entry unless there is a clinical suspicion of CNS involvement). Subjects with previously treated brain metastases may participate provided:

  * They are stable (without evidence of progression by imaging for at least four weeks and any neurologic symptoms have returned to baseline)
  * They have no evidence of new or enlarging brain metastases (confirmed by imaging within 28 days of the first dose of study drug)
  * They are not using steroids for at least 7 days before the first dose of study drug.

This exception does not include leptomeningeal metastases, which is excluded regardless of clinical stability.

* Has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days before study treatment.
* Has uncontrolled intercurrent illness including, but not limited to:

  * Uncontrolled infection
  * Disseminated intravascular coagulation
  * Psychiatric illness/social situations that would limit compliance with study requirements.
* Has known history positive status for human immunodeficiency virus or chronic active hepatitis B or hepatitis C (screening not required).
* Has any medical condition which in the opinion of the Investigator places the patient at an unacceptably high risk for toxicities.
* Use of prohibited medication within 7 days or 5 half-lives, whichever is shorter, prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Maximally Tolerated Dose (MTD) | Up to 21 days
  Starting at dose level 1, if 2/3 patients have a dose-limiting toxicity (DLT), the dose will be de-escalated to dose -1. If 0/3 patients experience a DLT, 3 patients will be treated at the next dose level. If DLT attributable to the treatment is experienced in 1/3 patients, three more patients (for a total of six patients) will be treated at that dose level. If no additional DLTs are observed at the expanded dose level (i.e. 1/6 with DLT), the dose will be escalated. Escalation will terminate as soon as two or more patients experience any DLT attributable to study drugs, at a given dose level. If de-escalation is necessary, 3 patients will be enrolled on the next lower dose cohort. If 1 or less DLTs is observed in this cohort, this will be the MTD.
Objective Response Rate (ORR) | Up to 2 years
  Objective response rate (ORR) by RECIST 1.1 criteria in patients treated with abexinostat in combination with (CPI) immune checkpoint inhibition in patients with prior primary or acquired resistance to prior CPI treatment.

SECONDARY OUTCOMES:
Immune-modified Objective response rate (ORR) | Up to 2 years
  Objective response rate (ORR) by iRECIST. The criteria are identical to those of RECIST 1.1 but have been adapted to account for instances where an increase in tumor burden, or the appearance of new lesions, does not reflect true tumor progression. Immuno response evaluation criteria in solid tumours (iRECIST) ORR requires the confirmation of progression and uses the terms unconfirmed progression (iUPD) and confirmed progression (iCPD).
Median Duration of Response (DoR) | Up to 2 years
  The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR), whichever is first recorded, until the first date that recurrent or progressive disease is objectively documented.
Median DoR per iRECIST | Up to 2 years
  The duration of overall response is measured from the time measurement criteria are met for CR (complete response) or PR (partial response), whichever is first recorded, until the first date that recurrent or progressive disease is objectively documented. The criteria are identical to those of RECIST 1.1 but have been adapted to account for instances where an increase in tumor burden, or the appearance of new lesions, does not reflect true tumor progression. iRECIST requires the confirmation of progression and uses the terms iUPD (unconfirmed progression) and iCPD (confirmed progression).
Median Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of initiation of study treatment to the date measurement criteria are first met for radiographic progressive disease (PD) or death from any cause, whichever occurs first.
Percentage of participants reporting treatment-related Adverse Events (AE) | Up to 2 years
  Percentages of participants experiencing adverse events by preferred term will be summarized by NCI-CTCAE version 5

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No